CLINICAL TRIAL: NCT03953391
Title: The Effect of Tea Breaks on Cerebrovascular Perfusion During Desk Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: REF-BEV-3235
Record Dates: First submitted 2019-04-24; First posted 2019-05-16 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Cerebrovascular Circulation; Affect
MeSH Terms: interventions — Tea; Water

STUDY DESIGN:
Intervention Model Description: Randomised, full cross-over study
Who Masked: Outcomes Assessor
Masking Description: Person doing the statistical analyses will blinded to the treatments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tea-water (Experimental): Tea before water
  Interventions: Other: Tea; Other: Water
- Water-tea (Experimental): Water before tea
  Interventions: Other: Tea; Other: Water

INTERVENTIONS:
Other: Tea — Subjects walk to a nearby area and prepare a cup of 150 ml tea once every hour. The tea is consumed whilst being seated at their desks.
Other: Water — 150 ml water is served to subjects once every hour. The water is consumed whilst being seated at their desks.

SUMMARY:
Sedentary behaviour of healthy subjects may have a detrimental impact on cerebral blood flow as well as cognitive measures related to mood and alertness. In this study we focus on the impact of leaving the desk to consume a cup of tea at regular intervals during a sedentary working day.

DETAILED DESCRIPTION:
Prolonged desk work has detrimental impact on cerebral blood flow as well as cognitive measures related to mood and alertness caused. These effects might be prevented by taking short breaks with physical activity. Usually, desk workers have short breaks during office times for either a visit to the restroom or to enjoy for a moment a (hot) drink. Consumption of tea has been associated with benefits related to attention, alertness, mood and creativity. This study focuses on the impact of physically leaving the desk to prepare and consume a cup of tea at regular intervals during a sedentary working day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, age at screening > 18 and < 60 years;
* BMI > 18 and < 30 kg/m2
* Apparently healthy
* Agreeing to be informed about medically relevant personal test-results by a physician
* Informed consent signed
* Sedentary working individuals (≥6 hours desk work per day, ≥4 days per week)

Exclusion Criteria:

* Reported physical exercise ≥4 hours per week
* Taking medication (including food supplements and traditional medicines) which may interfere with study measurements, as judged by the PI
* Reported participation in another nutritional or biomedical trial (involving an intervention of at least 1 week) 3 months before the screening or during the study
* Reported participation in night shift work 2 weeks prior to screening or during the study. Night work is defined as working between midnight and 6.00 a.m.
* Reported consumption of > 14 units (female subjects) and > 21 units (male subjects) alcoholic drinks in a typical week.
* Reported use of any nicotine containing products in the 6 months preceding the study and during the study itself.
* If female, is pregnant (or has been pregnant during the last < 3 months ago) or will be planning pregnancy during the study period.
* If female, is lactating or has been lactating in the 6 weeks before screening and/or during the study period.
* Reported weight loss/gain (> 10%) in the last 6 months before the study.
* Being an employee of Unilever or an employee or a student working in RISES LJMU that is directly involved in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Difference in cerebrovascular perfusion of tea versus water | Immediately before and immediately after each of the two 6-hour interventions. The 'before' results will be added to the mixed model as a covariate.
  Cerebrovascular perfusion measured as middle cerebral artery velocity

SECONDARY OUTCOMES:
Difference in cerebrovascular auto-regulation gain of tea versus water | Immediately before and immediately after each of the two 6-hour interventions. The 'before' results will be added to the mixed model as a covariate.
  Dynamic cerebrovascular autoregulation is assessed via squat-stand manoeuvres performed to elicit oscillations in blood pressure within the high-pass filter frequency range (<0.20 Hz) of the cerebrovascular. Squat-stand cycles are performed at 0.2 Hz (2.5-seconds squatting, followed by 2.5-seconds standing) and at 0.1 Hz (5-seconds squatting, followed by 5-seconds standing) for 5-minutes each, separated by a 5-minute rest.
  Transfer function analysis is conducted on the beat-to-beat blood pressure and middle cerebral artery blood flow velocity mean signals to produce values of gain (damping effect of Cerebrovascular autoregulation on the magnitude of blood pressure oscillations).
Difference in cerebrovascular auto-regulation phase of tea versus water | Immediately before and immediately after each of the two 6-hour interventions. The 'before' results will be added to the mixed model as a covariate.
  Dynamic cerebrovascular autoregulation is assessed via squat-stand manoeuvres performed to elicit oscillations in blood pressure within the high-pass filter frequency range (<0.20 Hz) of the cerebrovascular. Squat-stand cycles are performed at 0.2 Hz (2.5-seconds squatting, followed by 2.5-seconds standing) and at 0.1 Hz (5-seconds squatting, followed by 5-seconds standing) for 5-minutes each, separated by a 5-minute rest.
  Transfer function analysis is conducted on the beat-to-beat blood pressure and middle cerebral artery blood flow velocity mean signals to produce values of phase (temporal relationship between changes in blood pressure and middle cerebral artery blood flow velocity).
Difference in cerebrovascular auto-regulation coherence of tea versus water | Immediately before and immediately after each of the two 6-hour interventions. The 'before' results will be added to the mixed model as a covariate.
  Dynamic cerebrovascular auto-regulation is assessed via squat-stand manoeuvres performed to elicit oscillations in blood pressure within the high-pass filter frequency range (<0.20 Hz) of the cerebrovascular. Squat-stand cycles are performed at 0.2 Hz (2.5-seconds squatting, followed by 2.5-seconds standing) and at 0.1 Hz (5-seconds squatting, followed by 5-seconds standing) for 5-minutes each, separated by a 5-minute rest.
  Transfer function analysis is conducted on the beat-to-beat blood pressure and middle cerebral artery blood flow velocity mean signals to produce values of coherence (linearity of the relationship between the changes in middle cerebral artery blood flow velocity and blood pressure).

OTHER OUTCOMES:
Difference in PANAS of tea versus water | Immediately before and immediately after each of the two 6-hour interventions. The 'before' results will be added to the mixed model as a covariate.
  Positive and Negative Affect Schedule (PANAS) questionnaire consisting of a list of ten positive and ten negative feelings and emotions. Participants rate the extent to which they are feeling each emotion, on a scale from 1 (very slightly or not at all) to 5 (extremely).
Difference in Bond-Lader of tea versus water | Immediately before and immediately after each of the two 6-hour interventions. The 'before' results will be added to the mixed model as a covariate.
  Bond-Lader questionnaire: 16 adjective pairs with a 100mm line in between. Three sub-scales will be calculated: Alertness, Contentedness and Calmness.
Difference in affect of tea versus water | Before (0) and at 1, 2, 3, 4 and 5 hours during tea and water interventions. Both dimensions will be tested in a repeated measures linear mixed model. The treatment effect is the difference in the least square means of tea versus water.
  Affect grid. Two dimensional grid of 19x19 cells scoring pleasure and arousal

CONTACTS AND LOCATIONS:
Overall Officials: Dick Thijssen, prof, Principal Investigator — Liverpool John Moores University
Locations (1):
- John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No